CLINICAL TRIAL: NCT01683305
Title: Biomarker Breast Pap Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Silbiotech (Industry)
Responsible Party: Principal Investigator, Indira Poola, Ph.D, Principal Investigator, Silbiotech
Other Study IDs: Silbiotech:2012-01
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Tumors
Keywords: biomarker,; NAF; Subjects
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subjects who have no mammographically detectable tumors: This group will be evaluated for marker presence in NAF. no drugs administered
- Subjects who have non-cancerous growths: This group will be evaluated to study whether marker(s) detected in NAF are also expressed in non-cancerous tumors. No drugs administered
- subjects who have cancerous growths: In this group, any markers detected in NAF could also be detected in tumor tissues. No drugs administered.

SUMMARY:
This will be a Phase I study. During the Phase I study, our goals are: 1) screen a number of cancer biomarkers in Nipple Aspirate Fluid (NAF) from women who have no mammographically detectable tumors, and those who have detectable tumors, 2) identify all the detectable markers and 3) establish that biomarkers detected in NAF could also be detected in the biopsied tumor tissue that was removed for diagnostic purpose in subjects who have detectable tumors.

ELIGIBILITY:
Inclusion Criteria:

* Any female subject aged 18 years or older

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any woman age 18 or older
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)